CLINICAL TRIAL: NCT02907892
Title: Effect of Intra-operative Glove-changing During Cesarean Section on Post-op Complications:
Brief Title: Effect of Intra-operative Glove-changing During Cesarean Section on Post-op Complications: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1416
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-12

CONDITIONS: Wound Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard cesarean section surgical technique per surgeon preference
- Glove Change (Experimental): Cesarean section including changing of sterile surgical gloves immediately prior to abdominal closure
  Interventions: Procedure: Glove change

INTERVENTIONS:
Procedure: Glove change — Intra-operative changing of sterile surgical gloves immediately prior to abdominal closure during cesarean section
  Arms: Glove Change

SUMMARY:
A randomized controlled trial to determine whether changing of gloves by the surgical team during cesarean section may decrease post-operative infectious morbidity and wound complications

DETAILED DESCRIPTION:
This was a randomized, single-blind controlled trial of women who underwent cesarean section at Healthpartners Regions Hospital. Potential participants were identified during routine obstetrical care of singleton pregnancies at Regions Hospital, at the time that cesarean section was decided as the route of delivery by patient and provider. Patients were excluded if the cesarean section was performed emergently. Randomization occurred in the operating room during preparation for cesarean section; nursing staff drew a computer generated allocation card from a stack placed within an envelope in the room. Patients assigned to the control group underwent cesarean section with standard surgical technique at the discretion of the attending surgeon. Patients assigned to the glove change group underwent cesarean section in which the surgical team - surgeon, assistant, and scrub nurse - replaced their outer surgical gloves with a new sterile pair of gloves prior to abdominal closure. Abdominal closure was considered to begin with closure of the peritoneum, if performed, otherwise with closure of the abdominal fascia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with singleton pregnancy and shared decision making with provider resulting in plan for cesarean section

Exclusion Criteria:

* Severe immunocompromise (AIDS) or emergent nature of cesarean section

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Scrafford, MD, Principal Investigator — University of Minnesota
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Glove Change
Started | 277 | 276
Completed | 250 | 236
Not Completed | 27 | 40
Not completed — Lost to Follow-up | 27 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Glove Change | Total
Number analyzed (Participants) | 277 | 276 | 553
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.7 (5.3) | 30.6 (5.4) | 30.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 276 | 553
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 277 | 276 | 553

OUTCOME MEASURES:

1. Primary Outcome: Composite Wound Complication
Description: Occurence of at least one of the following: wound seroma, wound hematoma, wound infection, skin separation of at least 1cm, or other incisional separation or abnormality requiring a bedside procedure to fix
Time Frame: Within 8 weeks following cesarean section
Population: Participants with follow-up data (at least one postpartum visit within 8 weeks of delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Glove Change
Number analyzed (Participants) | 250 | 236
Participants | 34 | 15

ADVERSE EVENTS:
Arm/Group | Control | Glove Change
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/276
Other Adverse Events (participants affected / at risk) | 0/277 | 0/276

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes